CLINICAL TRIAL: NCT01930201
Title: Caudal Epidural Block for Postoperative Analgesia in Adolescents Following Major Hip Surgery.
Status: Completed | Type: Observational
Sponsor: David P. Martin (Other)
Responsible Party: Sponsor-Investigator, David P. Martin, Clinical Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB12-00842
Record Dates: First submitted 2013-07-09; First posted 2013-08-28 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Major Orthopedic Hip Surgery
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard general anesthesia: Patients receiving standard of care.
  Interventions: Other: General anesthesia
- Caudal Epidural Block: Patients receiving a caudal epidural block in addition to standard of care.
  Interventions: Procedure: Caudal epidural block; Other: General anesthesia

INTERVENTIONS:
Procedure: Caudal epidural block
  Groups: Caudal Epidural Block
Other: General anesthesia

SUMMARY:
This retrospective chart review will demonstrate the feasibility of performing caudal epidural blockade in adolescents undergoing major orthopedic hip surgery and provide information regarding the feasibility of this technique's use on a regular basis.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents that underwent major orthopedic hip surgery.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had major orthopedic hip surgery.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain | During 1st 24 hours post-op
  Assessing pain scores post-operatively.

SECONDARY OUTCOMES:
Pain medication requirement | During 1st 24 hours post-op
  Assessing amount of pain medication required.
Antiemetic medication requirement | During 1st 24 hours post-op
  Assessing need for antiemetic medications post-operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States